CLINICAL TRIAL: NCT02108587
Title: Staging of Upper Tract Urothelial Cancer With Optical Coherence Tomography
Brief Title: Optical Coherence Tomography in Staging Patients With Upper Tract Urothelial Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE11811; NCI-2014-00347 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 11811 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Kidney/Urinary Cancer
MeSH Terms: conditions — Urologic Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- optical coherence tomography for diagnosis (Experimental): Patients undergo optical coherence tomography over 10-15 minutes.
  Interventions: Device: optical coherence tomography

INTERVENTIONS:
Device: optical coherence tomography — Undergo optical coherence tomography

SUMMARY:
This clinical trial studies how well optical coherence tomography works in staging patients with upper-tract urothelial carcinomas. Staging describes the severity of a person's cancer based on the size and/or extent (reach) of the original (primary) tumor and whether or not cancer has spread in the body. It also helps the doctor plan the appropriate treatment. Optical coherence tomography is a procedure that uses infrared light waves to give three-dimensional pictures of structures inside tissues and organs. The pictures are made by a computer linked to the light source. Optical coherence tomography may be effective in staging patients with upper-tract urothelial carcinomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the feasibility and imaging ability of optical coherence tomography (OCT) to stage upper-tract urothelial carcinomas (UTUC).

OUTLINE:

Patients undergo optical coherence tomography over 10-15 minutes.

After completion of study, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiographic evidence of upper tract urothelial cancer by computed tomography (CT), magnetic resonance imaging (MRI) or intravenous pyelogram (IVP) in order to undergo this procedure
* Patient who will undergo standard of care clinical staging for UTUC
* Patient ability to read and comprehend the informed consent document

Exclusion Criteria:

* Patient who has a contraindication to endoscopy
* Patient who is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of optical coherence tomography (OCT) images in staging upper-tract urothelial carcinomas (UTUC) | Up to 3 months
  Feasibility defined as the ability to relate the features associated with cancerous tissues in pathohistological analysis to the features in OCT images

SECONDARY OUTCOMES:
Imaging Analysis | Up to 3 months
  Number of cancerous images with at least one feature different from normal pathology slide

CONTACTS AND LOCATIONS:
Overall Officials: Donald Bodner, MD, Principal Investigator — Case Comprehensive Cancer Center